CLINICAL TRIAL: NCT06315439
Title: Digital Confocal Microscopy for Real-time Diagnosis of Pancreatic Solid Lesion: a Multicentre Study
Brief Title: Digital Confocal Microscopy for Real-time Diagnosis of Pancreatic Solid Lesion
Acronym: Multi-RELAMI
Status: Completed | Type: Observational
Sponsor: Campus Bio-Medico University (Other)
Responsible Party: Principal Investigator, Francesco Maria Di Matteo, Head of Operative Digestive Endoscopy department, Campus Bio-Medico University
Other Study IDs: Multi-RELAMI
Record Dates: First submitted 2024-03-08; First posted 2024-03-18 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2024-03

CONDITIONS: Pancreas Adenocarcinoma; Endoscopic Ultrasound; Digital Pathology

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- pancreatic solid lesions
  Interventions: Procedure: Endoscopic ultrasound fine needle biopsy

INTERVENTIONS:
Procedure: Endoscopic ultrasound fine needle biopsy — EUS FNA/B for solid pancreatic lesions. After the FNA/FNB, the needle was removed from the EUS endoscope and the specimen obtained after the first needle pass was expelled and placed directly in a dedicated scaffold (Cytomatrix, UCS Diagnostics).
  a drop of ethanol was put on it and the liquid was drained away thanks to the porous structure of the matrix. This step was followed by the deposition of a drop of acridine-orange for 20" and a rapid washing with buffered saline. After that, the Cytomatrix was put on a dedicated microscopic slide and covered with a second slide before the introduction in the slot of the machine.
  The FCM VivaScope® 2500 (2500M-G4; VivaScope, Munich, Germany) was used for immediate imaging.

SUMMARY:
Endoscopic ultrasound-guided (EUS) tissue acquisition is the current standard of care for the diagnosis of pancreatic solid lesions but it is burdened by a non-negligible risk of non-diagnostic or inconclusive results.

Ex-vivo fluorescence confocal laser microscopy (FCM) with MAVIG VivaScope® 2500M-G4 could allow real time assessment of adequacy and diagnosis of the sample.

DETAILED DESCRIPTION:
Endoscopic ultrasound-guided (EUS) tissue acquisition is the current standard of care for the diagnosis of pancreatic solid lesions.

However, EUS-sampling is burdened by a non-negligible risk of non-diagnostic or inconclusive results, with an estimated negative predictive value not higher than 70-80%.

ROSE could improve the diagnostic yeld of this procedure. Data about the utility of rapid on-site evalutation (ROSE) are still controversial. Without ROSE, current guidelines suggest performance of three to four needle passes with an fine needle aspiration (FNA) needle or two to three passes with a fine needle biopsy (FNB) needle.

Potential drawbacks of ROSE are the considerable time commitment, costs and logistical and personnel issues that arise because of the "on demand" nature of these procedures with the need to have available technologists.

Ex-vivo fluorescence confocal laser microscopy (FCM) is an optical technology for rapid microscopic digital imaging of fresh unfixed biological specimens without any slide preparation.

FCM involves no damage or cell/tissue loss during the examination and the sample can subsequently be recovered and formalin-fixed and paraffin-embedded (FFPE) for permanent histology. FCM allows both cellular and architectural details to be visualized, similar to standard histological analysis of paraffin-embedded or frozen samples. With FCM, multimodal confocal microscopy using different laser sources and fusion images can generate optical plans similar to those from hematoxylin/eosin (H&E)- stained sections directly from native tissues.

Recently, the feasibility of FCM with MAVIG VivaScope® 2500M-G4 in EUS-FNB sample of pancreatic solid lesions has been investigated . This previous single-center study demonstrated good concordance between the FCM image-based evaluation and the final FFPE histology.

However in this first study, a single type of FNB needle was used for all the procedures and the pathologist involved was expert in digital pathology and in pancreatic disease. Therefore it might be not representative of the everyday clinical practice. In addition the first study was mainly focused on the adequacy assessment of the samples.

ELIGIBILITY:
Inclusion Criteria:

* pancreatic solid lesions

Exclusion Criteria:

* cystic lesions
* not suitable acoustic window for needle biopsy
* decline to give informed consent.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with solid pancreatic lesion will be enrolled
Sampling Method: Probability Sample
Enrollment: 78 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuracy | baseline
  To evaluate the accuracy of fluorescence confocal microscopy (FCM) for ex-vivo examination of samples obtained from EUS- FNA/B in pancreatic solid lesions to assess final diagnosis against final histological diagnosis.

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Policlinico Campus Bio Medico, Rome, ROMA, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Itoi T, Sofuni A, Itokawa F, Irisawa A, Khor CJ, Rerknimitr R. Current status of diagnostic endoscopic ultrasonography in the evaluation of pancreatic mass lesions. Dig Endosc. 2011 May;23 Suppl 1:17-21. doi: 10.1111/j.1443-1661.2011.01132.x. PMID 21535194
- [Background] Polkowski M, Jenssen C, Kaye P, Carrara S, Deprez P, Gines A, Fernandez-Esparrach G, Eisendrath P, Aithal GP, Arcidiacono P, Barthet M, Bastos P, Fornelli A, Napoleon B, Iglesias-Garcia J, Seicean A, Larghi A, Hassan C, van Hooft JE, Dumonceau JM. Technical aspects of endoscopic ultrasound (EUS)-guided sampling in gastroenterology: European Society of Gastrointestinal Endoscopy (ESGE) Technical Guideline - March 2017. Endoscopy. 2017 Oct;49(10):989-1006. doi: 10.1055/s-0043-119219. Epub 2017 Sep 12. PMID 28898917
- [Background] Facciorusso A, Wani S, Triantafyllou K, Tziatzios G, Cannizzaro R, Muscatiello N, Singh S. Comparative accuracy of needle sizes and designs for EUS tissue sampling of solid pancreatic masses: a network meta-analysis. Gastrointest Endosc. 2019 Dec;90(6):893-903.e7. doi: 10.1016/j.gie.2019.07.009. Epub 2019 Jul 13. PMID 31310744
- [Background] Gkolfakis P, Crino SF, Tziatzios G, Ramai D, Papaefthymiou A, Papanikolaou IS, Triantafyllou K, Arvanitakis M, Lisotti A, Fusaroli P, Mangiavillano B, Carrara S, Repici A, Hassan C, Facciorusso A. Comparative diagnostic performance of end-cutting fine-needle biopsy needles for EUS tissue sampling of solid pancreatic masses: a network meta-analysis. Gastrointest Endosc. 2022 Jun;95(6):1067-1077.e15. doi: 10.1016/j.gie.2022.01.019. Epub 2022 Feb 4. PMID 35124072
- [Background] Stigliano S, Crescenzi A, Taffon C, Covotta F, Hassan C, Antonelli G, Verri M, Biasutto D, Scarpa RM, Di Matteo FM. Role of fluorescence confocal microscopy for rapid evaluation of EUS fine-needle biopsy sampling in pancreatic solid lesions. Gastrointest Endosc. 2021 Sep;94(3):562-568.e1. doi: 10.1016/j.gie.2021.03.029. Epub 2021 Mar 31. PMID 33798539